CLINICAL TRIAL: NCT05044455
Title: Online Peer-Delivered Group CBT for Postpartum Depression
Brief Title: Online Peer-Delivered Group CBT for PPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Ryan Van Lieshout, MD, PhD, Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OnlinePeerCBT
Record Dates: First submitted 2021-09-02; First posted 2021-09-14 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Postpartum Depression
Keywords: CBT; Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial - Treatment group receives a 9 week on-line CBT treatment delivered by Peer facilitators as well as accessing treatment as usual for new mothers experiencing postpartum depression.
  Control Group accesses treatment as usual or typical treatment for new mothers in participant's communities and does not receive the CBT group.
Masking Description: Participants are assigned an identification number and data is de-identified during analysis phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Experimental, intervention (Experimental): The immediate intervention group will receive an online 9 week CBT intervention led by trained peers who have themselves recovered from postpartum depression. The CBT group will be two hours long, weekly and involves teaching and practice of core CBT skills. Core cognitive skills including thought records and cognitive restructuring are introduced and practiced from week 1. Behavioural techniques are introduced at week 2 and continue throughout the group, including behavioural activation, relaxation techniques, sleep strategies, exercise and goal setting. Each participant will receive a professionally design CBT manual to facilitate learning. Participants in the intervention group may also receive typical care or treatment as usual for new mothers.
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT)
- Arm 2: Control Group (No Intervention): The control group will receive treatment as usual (TAU) or typical care available for postpartum depression in participant's home communities, via participant's family doctor, mental health services, midwifery services, etc. Subjects in the control group will receive a list of resources where participants may seek treatment and will receive a monthly email encouraging them to seek treatment if symptoms worsen, including thoughts of self harm or harm to participant's child. Participants will also receive a copy of the Canadian Practice Guidelines for the treatment of PPD.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy (CBT) — A 9 week CBT group, 2 hours weekly, is delivered by trained Peer facilitators to mothers randomized to this arm.
  Arms: Arm 1: Experimental, intervention

SUMMARY:
Mothers and birthing parents (hereafter referred to as mothers) who have recovered from Postpartum Depression and are well now, receive training to teach a 9 week Cognitive Behavioural Therapy (CBT) treatment to mothers who are feeling depressed after giving birth in the last year. Eligible mothers are randomly assigned to one of two groups. Mothers in one group will receive a 9 week group CBT intervention delivered online by the trained Peer facilitators. Mothers in the other group will not receive the CBT group intervention and will continue to receive treatment as usual or regular care for new mothers.

Mothers in both groups will complete online questionnaires three times - when participants start the study, nine weeks later and six months after that. Mothers in the intervention group will also complete a few questionnaires once during the intervention and a satisfaction questionnaire at end of intervention. Participant information will help determine if the CBT treatment is helpful for postpartum depression.

DETAILED DESCRIPTION:
Mothers and birthing parents (hereafter referred to as mothers) who meet the eligibility criteria for the study (18+ years of age, with a baby under 12 months of age at recruitment, Edinburgh Postnatal Depression Scale (EPDS) score of 10 - 22 and living in Ontario are screened using the Mini International Neuropsychiatric Interview (MINI). Mothers free of bipolar, psychotic or current substance use disorders and borderline personality disorder are randomized 1:1 to the intervention (online 9 week peer-delivered CBT program) or control group (treatment as usual, TAU) after providing informed consent.

Participants in the Intervention Group receive a 9 week on-line CBT group (2 hrs weekly) delivered by Peer facilitators who have recovered from Postpartum Depression (PPD) and have been trained to deliver CBT. Participants may also continue to receive treatment as usual (medication, psychotherapy), or typical care, for new mothers from any source (healthcare providers, etc).

Participants in the Control Group do not receive the CBT group and are given a list of resources for mental health and postpartum depression supports and are also encouraged to seek treatment as usual or typical care for new mothers from any source. Participants will also receive follow up emails monthly with information about when to seek emergency treatment (if symptoms worsen, experience thoughts of self-harm or harm to the participant's baby).

All participants will receive personalized emails with links to participant's online questionnaires through REDCap at 3 time points (recruitment, nine weeks later and 6 months later). Participants in the intervention group will also complete questionnaires at one time point during the intervention and a satisfaction survey at end of intervention. The data from both groups will be examined to determine treatment effects and durability, respectively.

Peer facilitator fidelity to the CBT Model will be assessed using measures of adherence and competence and independently assessed by two raters.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* baby under 12 months of age at recruitment
* EPDS score 10 - 22
* lives in Ontario
* fluent in written/spoken English

Exclusion Criteria:

* Mothers and birthing parents who score positive on the MINI subsections of bipolar, psychotic, current substance abuse disorders and/or borderline personality disorder

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers and birthing parents who have given birth within 12 months
Enrollment: 191 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | 9 weeks
  The Edinburgh Postnatal Depression Scale (EPDS) is the 10-item gold standard measure of PPD. Total scores range from 0-30 with higher scores indicating worse depressive symptoms.. A score ≥13 is consistent with PPD and changes in scores >4 are accepted as being indicative of clinically significant change
Edinburgh Postnatal Depression Scale (EPDS) | 6 months
  The Edinburgh Postnatal Depression Scale (EPDS) is the 10-item gold standard measure of PPD. Total scores range from 0-30 with higher scores indicating worse depressive symptoms.. A score ≥13 is consistent with PPD and changes in scores >4 are accepted as being indicative of clinically significant change
MINI International Neuropsychiatric Interview | 9 weeks
  A brief structured interview for the major Axis 1 psychiatric disorders in the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM 5) . Major Depressive Disorder Module to determine if participants meet diagnostic criteria for PPD at 9 weeks
MINI International Neuropsychiatric Interview | 6 months
  A brief structured interview for the major Axis 1 psychiatric disorders in the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM 5). Major Depressive Disorder Module to determine if participants meet diagnostic criteria for PPD at six months

SECONDARY OUTCOMES:
GAD-7 | 9 weeks
  The Generalized Anxiety Disorder 7-Item Scale (GAD-7) (32) is a self-report scale that taps generalized anxiety disorder, the most common comorbidity of PPD. Items are scored on a 4-point scale from 0 to 3, with a higher score indicating an increased risk of GAD. A cutoff of ≥11 defines clinically important levels of anxiety symptoms.
GAD-7 | 6 months
  The Generalized Anxiety Disorder 7-Item Scale (GAD-7) (32) is a self-report scale that taps generalized anxiety disorder, the most common comorbidity of PPD. Items are scored on a 4-point scale from 0 to 3, with a higher score indicating an increased risk of GAD. A cutoff of ≥11 defines clinically important levels of anxiety symptoms.
Multidimensional Scale of Perceived Social Support (MSPSS) | 9 weeks
  A 12-item scale designed to measure perceived social support from three sources: (1) family, (2) friends and (3) significant other. Items are scored on a 7-point scale, and total scores range from 12-84 with higher scores indicating a higher level of perceived social support. A score of 12-35 indicates low perceived social support, 36-60 indicates medium perceived social support and 61-84 indicates high perceived social support.
Multidimensional Scale of Perceived Social Support (MSPSS) | 6 months
  A 12-item scale designed to measure perceived social support from three sources: (1) family, (2) friends and (3) significant other. Items are scored on a 7-point scale, and total scores range from 12-84 with higher scores indicating a higher level of perceived social support. A score of 12-35 indicates low perceived social support, 36-60 indicates medium perceived social support and 61-84 indicates high perceived social support.
The Postpartum Bonding Questionnaire (PBQ) | 9 weeks
  The Postpartum Bonding Questionnaire (PBQ) is a 25-item maternal-report measure that assesses four aspects of maternal-infant relations: (1) bonding, (2) rejection and anger towards the infant, (3) infant-focused anxiety and (4) incipient abuse. Subscales 1-3 will be explored as a continuous outcome using subscale total score. Each item is scored on a scale of 0-5, with higher scores suggestive of more problems. Mother-infant bonding will be measured as a continuous and dichotomous outcome, using cut-off scores for each subscale indicating bonding disorders. Cutoff values of 12 for the bonding subscale, 17 for rejection and anger, and 10 for infant-focused anxiety have been proposed to define bonding disorders in each category.
The Postpartum Bonding Questionnaire (PBQ) | 6 months
  The Postpartum Bonding Questionnaire (PBQ) is a 25-item maternal-report measure that assesses four aspects of maternal-infant relations: (1) bonding, (2) rejection and anger towards the infant, (3) infant-focused anxiety and (4) incipient abuse. Subscales 1-3 will be explored as a continuous outcome using subscale total score. Each item is scored on a scale of 0-5, with higher scores suggestive of more problems. Mother-infant bonding will be measured as a continuous and dichotomous outcome, using cut-off scores for each subscale indicating bonding disorders. Cutoff values of 12 for the bonding subscale, 17 for rejection and anger, and 10 for infant-focused anxiety have been proposed to define bonding disorders in each category.
Infant Behavior Questionnaire-Revised Very Short Form (IBQ-R) | 9 weeks
  The Infant Behaviour Questionnaire-Revised (Very Short Form) (IBQR) is a parent-report measure of infant temperament. The IBQ-R (Very Short Form) consists of 37 items answered on a 7-point scale (1-7) and assesses 3 factors: Positive Affectivity/Surgency with 13 items, Negative Emotionality with 12 items, and Orienting/Regulatory Capacity with 12 items; higher scores indicate greater alignment with the domain.
Infant Behavior Questionnaire-Revised Very Short Form (IBQ-R) | 6 months
  The Infant Behaviour Questionnaire-Revised (Very Short Form) (IBQR) is a parent-report measure of infant temperament. The IBQ-R (Very Short Form) consists of 37 items answered on a 7-point scale (1-7) and assesses 3 factors: Positive Affectivity/Surgency with 13 items, Negative Emotionality with 12 items, and Orienting/Regulatory Capacity with 12 items; higher scores indicate greater alignment with the domain.
EQ-5D-5L | 9 weeks
  A utility-based health-related quality of life self-report instrument consisting of five questions covering mobility, self-care, usual activities, pain/discomfort and depression/anxiety. Quality of Life will be calculated using the Canadian scoring algorithm by multiplying the health utility for the corresponding time period (ie. area under the curve approach).
EQ-5D-5L | 6 months
  A utility-based health-related quality of life self-report instrument consisting of five questions covering mobility, self-care, usual activities, pain/discomfort and depression/anxiety. Quality of Life will be calculated using the Canadian scoring algorithm by multiplying the health utility for the corresponding time period (ie. area under the curve approach).
Healthcare Resource Utilization Questionnaire | 9 weeks
  Healthcare resource utilization data will be collected using a questionnaire used in prior work and adapted for the postpartum period based on the Canadian Community Health Survey and Service Use and Resources Form. Participants will be asked to provide information on health care resource use including diagnoses and procedures, medications, hospital stays, physician and ER visits and the use of all other services (including those relating to mental health). The investigators will measure resources consumed from the perspective of public health care payer and corresponding unit costs will be calculated using provincial billing rates.
Healthcare Resource Utilization Questionnaire | 6 months
  Healthcare resource utilization data will be collected using a questionnaire used in prior work and adapted for the postpartum period based on the Canadian Community Health Survey and Service Use and Resources Form. Participants will be asked to provide information on health care resource use including diagnoses and procedures, medications, hospital stays, physician and ER visits and the use of all other services (including those relating to mental health). The investigators will measure resources consumed from the perspective of public health care payer and corresponding unit costs will be calculated using provincial billing rates.

OTHER OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | 9 weeks
  Intervention participants only. An 8-item scale that measures and assesses consumer satisfaction with health and human services. Items are scored on a 4-point scale and total scores range from 8-32, with higher scores indicating greater satisfaction.
CBT Skills Questionnaire (CBTSQ) | 4 weeks
  Intervention participants only. A 16-item maternal-report measure designed to assess cognitive and behavioural skills acquisition. Each item is scored on a 5-point scale, and total scores range from 16-80. Higher cognitive restructuring and behavioural activation scores predict reduction of overall psychiatric symptoms and depression.
CBT Skills Questionnaire (CBTSQ) | 9 weeks
  Intervention participants only. A 16-item maternal-report measure designed to assess cognitive and behavioural skills acquisition. Each item is scored on a 5-point scale, and total scores range from 16-80. Higher cognitive restructuring and behavioural activation scores predict reduction of overall psychiatric symptoms and depression.
Working Alliance Inventory (WAI-SR) | 4 weeks
  Intervention participants only. A 12-item maternal-report measure that assesses three aspects of therapeutic alliance:(1) agreement on the tasks of therapy, (2) agreement on the goals of therapy and (3) development of an affective bond. Items are rated on a 5-point scale, and total scores range from 12-60 with higher scores indicating a better therapeutic alliance.
Working Alliance Inventory (WAI-SR) | 9 weeks
  Intervention participants only. A 12-item maternal-report measure that assesses three aspects of therapeutic alliance:(1) agreement on the tasks of therapy, (2) agreement on the goals of therapy and (3) development of an affective bond. Items are rated on a 5-point scale, and total scores range from 12-60 with higher scores indicating a better therapeutic alliance.
Peer Support Integrity, Quality and Impact Survey (PSIQI) | 4 weeks
  Intervention participants only. A 4-scale maternal-report measure used to evaluate therapy quality. Subscale 1 will be explored which includes 17 statements about possible actions and behaviours of a peer support worker. Items are scored on a 5 point-scale, with "not applicable" available as a sixth option (this score is excluded when total score is calculated). The score range for Subscale 1 is 17-85 with a higher score indicating more positive feelings about the therapist's integrity.
Peer Support Integrity, Quality and Impact Survey (PSIQI) | 9 weeks
  Intervention participants only. A 4-scale maternal-report measure used to evaluate therapy quality. Subscale 1 will be explored which includes 17 statements about possible actions and behaviours of a peer support worker. Items are scored on a 5 point-scale, with "not applicable" available as a sixth option (this score is excluded when total score is calculated). The score range for Subscale 1 is 17-85 with a higher score indicating more positive feelings about the therapist's integrity.
Therapeutic Factors Inventory 8 (TFI-8) | 4 weeks
  An 8-item self-report measure that assesses individuals' perception of four therapeutic factors in group settings: (1) instillation of hope, (2) secure emotional expression, (3) awareness of relational impact, and (4) social learning.
Therapeutic Factors Inventory 8 (TFI-8) | 9 weeks
  An 8-item self-report measure that assesses individuals' perception of four therapeutic factors in group settings: (1) instillation of hope, (2) secure emotional expression, (3) awareness of relational impact, and (4) social learning.
Adherence Checklist | Weekly, weeks 1 through 9 of intervention
  9 individual checklists that measure the degree to which a peer leader is consistent with the intervention manual when applying techniques. The nine sessions vary in content, so this scale consists of different items for each session and assesses topics including agenda setting, content delivery, and homework review. Individual items are rated on a 3-4-point Likert scale ranging from 0 (not covered at all) to 3 (or 4) thorough coverage. Total adherence scores range from 15 (session 4, 6, 9) to 31 (session 1). These checklists are used by the peers, expert therapist (psychiatrist) and a graduate student
Competence Checklist | Weekly, weeks 1 through 9 of intervention
  This one checklist measures the level of skill and judgement that a peer leader demonstrates when delivering the intervention. This scale assesses structure and use of time, genuineness, empathy, collaboration, guided discovery, group participation, and eliciting emotional expression. Competence scores range from 0-42 with a higher score indicating greater competence.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Van Lieshout, MD PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Crick K, Al Sayah F, Ohinmaa A, Johnson JA. Responsiveness of the anxiety/depression dimension of the 3- and 5-level versions of the EQ-5D in assessing mental health. Qual Life Res. 2018 Jun;27(6):1625-1633. doi: 10.1007/s11136-018-1828-1. Epub 2018 Mar 7. PMID 29516342
- [Background] Xie F, Pullenayegum E, Gaebel K, Bansback N, Bryan S, Ohinmaa A, Poissant L, Johnson JA; Canadian EQ-5D-5L Valuation Study Group. A Time Trade-off-derived Value Set of the EQ-5D-5L for Canada. Med Care. 2016 Jan;54(1):98-105. doi: 10.1097/MLR.0000000000000447. PMID 26492214
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Loyd BH, Abidin RR. Revision of the Parenting Stress Index. J Pediatr Psychol. 1985 Jun;10(2):169-77. doi: 10.1093/jpepsy/10.2.169. No abstract available. PMID 4020601
- [Background] Brockington IF, Fraser C, Wilson D. The Postpartum Bonding Questionnaire: a validation. Arch Womens Ment Health. 2006 Sep;9(5):233-42. doi: 10.1007/s00737-006-0132-1. Epub 2006 May 4. PMID 16673041
- [Background] Putnam SP, Helbig AL, Gartstein MA, Rothbart MK, Leerkes E. Development and assessment of short and very short forms of the infant behavior questionnaire-revised. J Pers Assess. 2014;96(4):445-58. doi: 10.1080/00223891.2013.841171. Epub 2013 Nov 9. PMID 24206185
- [Background] Chiara G, Eva G, Elisa M, et al. Psychometrical properties of the Dyadic Adjustment Scale for measurement of marital quality with Italian couples. Procedia-Social and Behavioral Sciences. 2014;127:499-503. doi:10.1016/j.sbspro.2014.03.298
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Hepner KA, Howard S, Paddock SM, et al. A Fidelity Coding guide for a Group Cognitive Behavioral Therapy for Depression: RAND Corporation. 2011
- [Background] Jacob KL, Christopher MS, Neuhaus EC. Development and validation of the cognitive-behavioral therapy skills questionnaire. Behav Modif. 2011 Nov;35(6):595-618. doi: 10.1177/0145445511419254. Epub 2011 Sep 5. PMID 21893554
- [Background] Munder T, Wilmers F, Leonhart R, Linster HW, Barth J. Working Alliance Inventory-Short Revised (WAI-SR): psychometric properties in outpatients and inpatients. Clin Psychol Psychother. 2010 May-Jun;17(3):231-9. doi: 10.1002/cpp.658. PMID 20013760
- [Background] Peer Support Integrity, Quality and Impact Survey, 1.1 ed. Centre for Innovation in Peer Support. Hamilton, ON, Canada. April. 2019
- [Background] Matsubara C, Green J, Astorga LT, Daya EL, Jervoso HC, Gonzaga EM, Jimba M. Reliability tests and validation tests of the client satisfaction questionnaire (CSQ-8) as an index of satisfaction with childbirth-related care among Filipino women. BMC Pregnancy Childbirth. 2013 Dec 17;13:235. doi: 10.1186/1471-2393-13-235. PMID 24341288